CLINICAL TRIAL: NCT02657642
Title: The OMAGE (Optimization of Medication in AGEd) Transitional Care-Pathway: Impact on Readmissions
Acronym: OMAGE-P
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 15-086
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Ageing
Keywords: drug related problems, elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1 (exposed): cohort 1: patients who will receive the OMAGE-P transitional care in geriatric or internal medicine departement of the Eaubonne Hospital
- Cohort 2 (non exposed): Cohort 2: : patients included in the usual care arm of the OMAGE RCT study in 2007-2008

SUMMARY:
Background : The transitional care OMAGE-P combines three best practices recommendations from the French National Authority for Health (HAS) (i) a comprehensive review of diagnosis and treatments (ii) a standardized medical report and (iii)a patient education program specifically designed for older people with multiple chronic conditions and polypharmacy. This transitional care is implemented in a pilot general hospital with the support of French ministry of Health and Regional Agency for Health of Ile de France . The aim of the study is to assess the impact of the OMAGE P transitional care on the readmissions of non demented older people aged 75 years and over within the 3 months following their discharge to home and its cost-effectiveness .

Study Population: non demented people aged 75 years and over admitted in emergency (ie via an emergency department ) in the participating units

Study design:

Observational prospective monocentric non randomized comparative study Exposed patients: eligible patients admitted in participating units and who does not oppose to the collection of his personal data. The hospital physician in charge will conduct the comprehensive review of diagnosis and treatments and will do the standardized medical report. Patient education program will be conduct by the hospital physician and the OMAGE nurse during the hospitalization (two sequences) and during 2 to 4 home visits in the month following patient 's discharge from hospital.

Non exposed patients: eligible patients from the usual care arm of the RCT OMAGE. To ensure that risk for emergency readmissions is not different between exposed and non exposed , the rate of emergency readmissions of non exposed group will be compared with the one of eligible patient admitted in the participating units in 2013 and 2014.

Setting: General hospital of Eaubonne : geriatric department (acute geriatric unit, rehabilitation unit , geriatric mobile unit ) and internal medicine department Number of subjects to be included: 484 (242 in each arm). The data for the 242 non exposed patients are still available, 242 patients has to be included in the exposed group

DETAILED DESCRIPTION:
Background : The transitional care OMAGE-P combines three best practices recommendations from the French National Authority for Health (HAS) (i) a comprehensive review of diagnosis and treatments (ii) a standardized medical report and (iii)a patient education program specifically designed for older people with multiple chronic conditions and polypharmacy. This transitional care is implemented in a pilot general hospital with the support of French ministry of Health and Regional Agency for Health of Ile de France .The aim of the study is to assess the impact of the OMAGE P transitional care on the readmissions of non demented older people aged 75 years and over within the 3 months following their discharge to home and its cost-effectiveness Study Population: non demented people aged 75 years and over admitted in emergency (ie via an emergency department ) in the participating units

Study design:

Observational prospective monocentric non randomized comparative study Exposed patients: eligible patients admitted in participating units and who does not oppose to the collection of his personal data. The hospital physician in charge will conduct the comprehensive review of diagnosis and treatments and will do the standardized medical report. Patient education program will be conduct by the hospital physician and the OMAGE nurse during the hospitalization (two sequences) and during 2 to 4 home visits in the month following patient 's discharge from hospital.

Non exposed patients: eligible patients from the usual care arm of the RCT OMAGE (Legrain et al, JAGS, 2011). To ensure that risk for emergency readmissions is not different between exposed and non exposed , the rate of emergency readmissions of non exposed group will be compared with the one of eligible patient admitted in the participating units in 2013 and 2014.

Setting: General hospital of Eaubonne : geriatric department (acute geriatric unit, rehabilitation unit , geriatric mobile unit ) and internal medicine department The OMAGE-P transitional care: this transitional care is derived from the OMAGE intervention, which has proved to be associated with a significant reduction of readmitted patient 3 month after their discharge from acute geriatric unit (, 20.2% of Intervention group participants had been readmitted on an emergency basis, compared with 28.4% of control group participants, P = .01, RRR = 28.9%, 95% CI = 6.0-51.5%, Legrain et al JAGS 2011). The OMAGE -P transitional care consisted in (i) a comprehensive review of diagnosis and treatments, performed by hospital physician. The physician of participating units have been training to this medical review using a simple tool derived from a HAS program for the optimization of prescription in elderly. This tool consists in a table confronting patient's health problems and its treatments . This review necessitate an in depth treatments history (performed by physician in collaboration with usual patient's pharmacist ), a collaboration with general practitioner and an assesment of patient's problems regarding drug management (including adherence, self-medication ..etc) performed by the OMAGE nurse.

(ii) a standardized medical report. This report relies on the HAS recommendations regarding medical report which include notably a table indicating drugs at admission, drugs at discharge and reasons for modifications.

(iii) a patient education program specifically designed for older people with multiple chronic conditions and polypharmacy . This program aimed to promote the participant as active partners in care by assessing the participants' health priorities (preferences, values, and treatment burden) and strengthening participants' ability to better manage their own follow-up. It consists in two sequences at hospital (educational assessment by OMAGE nurse and sequence about links between patient's health problems by hospital physician) and 2 to 4 sequences during home visits by OMAGE nurse about red flags and situations at risk for patient's health, drug management and nutrition and physical activities adapted to patient's health. The OMAGE nurse performs this visits in close collaboration with GP and usual health professionals implicate din patient's care.

Statistical analysis: intention to treat analysis . Our hypothesis, based on the results of the OMAGE RCT, is that the OMAGE P transitional care is associated with a reduction in 3-month emergency readmissions from 30% to 20%. To detect such reduction with 80% power and an alpha risk of 5%, 242 participants are required per arm.

ELIGIBILITY:
Inclusion criteria:

* Aged 75 years and over
* Admitted in emergency (ie via an emergency unit)
* Living in a pre-defined territory (surroundings of the Eaubonne hospital)
* Not living in nursing home or no anticipated discharge in nursing home
* Not suffering from dementia
* Not receiving palliative care

Non inclusion criteria

* Patient's Opposition to collection of his personal data
* Previous participation in the OMAGE-P study,
* Inclusion in another therapeutic trial,
* Not speaking french,
* Impossible to follow up
* Absence of any health insurance (as required by French law on clinical research).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: non demented older people aged 75 years and over admitted in emergency in medical units living in community
Sampling Method: Non-Probability Sample
Enrollment: 484 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of days alive and without emergency readmissions | up to 6 months after hospital discharge
  Emergency visits and mortality will be assessed in the same way as readmissions. Vital status of patients lost to follow-up will be assessed by By contacting the town hall of the born municipality. Drug related readmissions will be assessed by an expert committee who will adjudicate whether readmissions are drug related. The adjudication process will rely on medical hospital discharge reports for each readmission (and additional data on request, such as medical records, biological results, electrocardiographs) and will follow a standardized guide. Disagreements will be resolved by consensus between the experts. The items in the adjudication guide will include : cause(s) for readmission, ﬁnal diagnosis or diagnoses, imputability of drug related problems (ADRs, adherence problems, underuse) in the readmission. Death during readmission will be systematically adjudicated

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Legrain, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No